CLINICAL TRIAL: NCT06788483
Title: The Effects of Self-regulated Flipped Classroom Strategy on Nursing Students' Self-regulated Learning Abilities, Self-efficacy and Nursing Skill Performance: a Randomized Controlled Study
Brief Title: Self-regulated Flipped Classroom Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Miao-Yi Chen, National Defense Medical Center, Taiwan, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CGUST
Record Dates: First submitted 2025-01-15; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Self-regulated Flipped Classroom Strategy; Self-Efficacy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): An self-regulated flipped classroom strategy
  Interventions: Behavioral: An self-regulated flipped classroom strategy
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: An self-regulated flipped classroom strategy — The self-regulated flipped classroom strategy was developed based on the self-regulated learning theory (Zimmerman, 2002) and the flipped classroom model (Bishop & Verleger, 2013).
  Arms: Intervention group

SUMMARY:
To examine the effect of a self-regulated flipped classroom strategy on nursing students' self-regulation abilities and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* (1) second-year undergraduate nursing students (2) students taking the Adult Nursing course this semesterand (3) willingness to participate in the study.

Exclusion Criteria:

* (1) having to quit school.

Ages: 18 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
self-regulated learning | 4 months
  self-regulated learning scale

SECONDARY OUTCOMES:
self-efficacy | 4 months
  Self-efficacy Scale (SES)

CONTACTS AND LOCATIONS:
Locations (1):
- Ting-Yu, Chen, Chiayi County, Puzi City, Taiwan

IPD SHARING:
Plan to Share IPD: No